CLINICAL TRIAL: NCT03348774
Title: Scrutinizing the Heterogeneity of Systemic Lupus Erythematosus: Defining Phenotypes
Brief Title: Scrutinizing the Heterogeneity of SLE: Defining Phenotypes
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Health Network, Toronto (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Murray B Urowitz, MD FRCP(C), Priniple Investigator, University Health Network, Toronto
Other Study IDs: 17-5083
Record Dates: First submitted 2017-07-24; First posted 2017-11-21 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Disease Course
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SLE disease course is characterized by unpredictable relapses and remissions in the majority of patients. However, in a small proportion (approximately 5%), SLE presents with a monophasic pattern, meaning that these patients have active disease before and immediately after diagnosis and after some time they achieve prolonged remission (for 12 years on average). Interestingly, about half of these patients do so and require no medications. On the other end of the clinical spectrum, approximately 50% of the patients demonstrate persistent disease activity and usually have the highest risk for developing co-morbidities and irreversible damage. A major goal of clinical research in SLE is to improve disease management based on disease course. By better characterizing SLE disease course we hope to better identify patients early in the disease course for targeted therapies to prevent and or reduce future SLE complications.

The overall objective of our project is to define distinct phenotypes of SLE based on disease course, clinical features, pathogenic mechanisms, genetic factors and relevant biomarkers.

DETAILED DESCRIPTION:
Specific aims of this study are:

1. To test the clinical impression of the disease courses by modeling the course of the disease in each of three sub-populations of patients where it is anticipated that one sub-population will experience relapsing and remitting disease activity, one will experience persistently active disease and another will exhibit a monophasic pattern.
2. To develop predictive models for group membership to enhance the accuracy of prognosis.
3. To test these models in the inception cohort of SLE patients within the Toronto Lupus Cohort.

Study Design: Retrospective longitudinal observational cohort

Patients will be categorised into three disease courses:

I. Relapsing-remitting II. Persistently active III. Monophasic Relapsing/remitting is defined as periods of disease activity SLEDAI-2K of 4 or more, (but if only 4 cannot be from serology alone) less than 50% of the time alternating with periods of inactivity (SLEDAI-2K <4) over the course of follow-up.

Persistently active disease is defined as SLEDAI-2K of 4 or more, (but if only 4 cannot be from serology alone), in greater than 80% of the visits, or no 2 consecutive visits with SLEDAI-2K < 4.

Monophasic course is defined as disease activity SLEDAI-2K of 4 or more, (but if only 4 cannot be from serology alone) for an initial period of less than 3 years followed by resolution and inactive disease (SLEDAI-2K of 0 excluding serology) for at least 5 years.

Clinical and laboratory characteristics, therapies and outcomes for each subgroup will be described. Identification of all clinical and laboratory features of lupus contained in the CRF will be compared for each group, as well as the medications prescribed.

ELIGIBILITY:
Inclusion Criteria:

Patients enrolled in the study for aims 1 and 2 must meet the following inclusion criteria:

1. ≥4 American College of Rheumatology (ACR) criteria or 3 ACR criteria plus a typical histological lesion of SLE on renal or skin biopsy.
2. Patients must have a minimum of 2 assessment visits.

Patients enrolled in the study for aim 3 must meet the following criteria:

1. Must be inception patients seen within one year of diagnosis of SLE
2. ≥4 American College of Rheumatology (ACR) criteria or 3 ACR criteria plus a typical histological lesion of SLE on renal or skin biopsy.
3. Patients must have a minimum of 6 assessment visits to ensure categorization into one of the disease courses derived in aims 1 and 2

Exclusion Criteria:

1. Patients who have not had 2 assessment visits for aims 1 and 2
2. Patients who have not had 6 assessments for aim 3.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with SLE have been followed prospectively at the University of Toronto Lupus Clinic since 1970. All patients ≥4 or more of the 1997 ACR criteria for SLE, or have 3 criteria and a typical lesion of SLE on renal or skin biopsy. Patients are evaluated at 2-6 month intervals according to a standard protocol which includes a detailed clinical history, physical examination, and laboratory evaluation . It includes all information necessary to calculate disease activity and damage indices, as well as comorbidities. Disease activity is assessed by the SLE Disease Activity Index 2000 (SLEDAI-2K) , and accumulated damage by the SLICC/ACR damage index (SDI) .
  To date there are 1767 patients with 2 or more visits registered in the Lupus Clinic Database, with 43079 assessments recorded. Their characteristics are shown in Table 1.
Sampling Method: Probability Sample
Enrollment: 950 (Estimated)
Dates: Start 2017-02-09 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
Disease Course Patterns | 6 months
  All 49,000 visits within the Toronto Lupus Cohort will be probed for patterns of disease activity using SLEDAI-2K measurements on each assessment. A finite mixture model will be fitted to the data to accommodate for three sub-populations of patients. Disease course for each sub-populations will be defined in terms of multistate model where the states reflected meaningfully different degrees of disease activity as measured by the SLEDAI-2K scores.

CONTACTS AND LOCATIONS:
Overall Officials: Murray Urowitz, Principal Investigator — University Health Network and University of Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No IPD data will be shared with other researchers